CLINICAL TRIAL: NCT01045915
Title: Safety and Efficacy of Intratumoural Electrotransfer of Plasmid AMEP in Patients Suffering From Advanced or Metastatic Melanoma: an Open Phase 1 Trial
Brief Title: Safety and Efficacy Study of Electrotransfer of Plasmid AMEP to Treat Advanced or Metastatic Melanoma
Acronym: AMEP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been halted due to the low enrolment rate.
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA2009/15/01; 2009-013042-88 (Registry Identifier: EudraCT number)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2012-05

CONDITIONS: Melanoma
Keywords: Stage IIIB, stage IIIC or stage IV melanoma; Progressive melanoma not responding to previous treatments
MeSH Terms: conditions — Melanoma | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plasmid AMEP electrotransfer (Experimental)
  Interventions: Biological: naked DNA coding for protein AMEP

INTERVENTIONS:
Biological: naked DNA coding for protein AMEP — 2 injections 1 week interval of 4 increasing doses of plasmid with electrotransfer
  Other Names: electrotransfer; electroporation

SUMMARY:
The objective of the present trial is to evaluate the local and general safety of the intratumoural electrotransfer of increasing doses of Plasmid AMEP in patients suffering from advanced or metastatic melanoma and to identify doses that could be effective on cutaneous lesions in man.

DETAILED DESCRIPTION:
In this open, multicentre, dose escalation study, successive cohorts of 3 patients suffering from advanced or metastatic melanoma will be electrotransferred increasing doses of Plasmid AMEP into cutaneous melanoma lesions in 2 divided doses at one week interval.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-breast feeding female;
2. Aged between 18 and 75 years;
3. Stage IIIB, stage IIIC or stage IV melanoma with:

   * At least 2 cutaneous or subcutaneous non necrotic accessible tumours;
   * Tumour size of 1 to 1.5 cm diameter;
   * No minimum distance between the 2 selected lesions;
4. Progressive melanoma not responding to previous treatments or patients refusing other therapies;
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
6. For women of child-bearing age: effective contraception method (oral contraception or intra-uterine device) used for more than 2 months before the 1st administration and to be maintained for 3 months after the last administration of Plasmid AMEP;
7. Having given a written informed consent.

Exclusion Criteria:

1. Patients who can benefit from other melanoma treatments including surgery;
2. Significant cardiac arrhythmias, electronic pacemakers, defibrillators, or any implanted electronic device;
3. Recent (less than 6 months) acute vascular diseases (stroke, MI…);
4. Advanced peripheral arterial diseases, venous ulcers, or scleroderma;
5. History or treatment of seizures within the last 5 years;
6. Clinically significant abnormality at pre-study full physical examination;
7. Any clinically significant ECG abnormalities;
8. Prior systemic therapy or any other antineoplastic treatments within the last 4 weeks, radiotherapy or surgery unrelated to the fields in question are allowed;
9. Abnormal renal function (creatinine plasma level > ULN);
10. Abnormal liver function tests (any of the following):

    * PT < 70%, ASAT, ALAT, alkaline phosphatases, GGT and/or total bilirubin > ULN in the absence of liver metastasis;
    * PT < 70%, ASAT, ALAT > 2 ULN, alkaline phosphatases > 1.5 ULN, GGT > 5 ULN and/or total bilirubin > 3 ULN in the case of liver metastases;
11. Abnormal bone marrow function: haemoglobin < 10g/dL, WBC < 3.109 /L and/or platelet count < 100.103 /L;
12. Clinically significant abnormality in pre-study laboratory tests;
13. Evidence of significant active infection (e.g., pneumonia, wound abscess, etc);
14. Intractable coagulopathy;
15. Any significant disease, including psychiatric and dermatology diseases that may affect the proper evaluation of efficacy or safety;
16. Patients who had participated in another clinical trial in the last 30 days prior to enrolment in the present clinical trial;
17. Patients unwilling or unable to comply with protocol requirements and scheduled visits.

Note: patients with brain metastases, or waiting for other therapies (i.e. isolated limb perfusion) may be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determination of Dose Limiting Toxicity defined as any grade 4 clinical, biological or any life-threatening ECG event occurring during the 9 weeks following treatment | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ATTALI Pierre, MD, Study Director — BioAlliance Pharma
Locations (3):
- Copenhagen University Hospital Herlev, Herlev, Denmark
- Gustave Roussy Institute, Le Kremlin-Bicêtre, France
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

REFERENCES:
- See also: Gene electrotransfer of plasmid antiangiogenic metargidin peptide (AMEP) in disseminated melanoma: safety and efficacy results of a phase I first-in-man study. — http://www.ncbi.nlm.nih.gov/pubmed/23980876